CLINICAL TRIAL: NCT03648970
Title: Pravastatin to Prevent Preeclampsia and Reduce Maternal-Neonatal Mortality and Morbidity in High Risk Preeclampsia Patients
Brief Title: Indonesia Pravastatin to Prevent Preeclampsia Study
Acronym: INOVASIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Muhammad Ilham Aldika Akbar, MD, OBGYN, Principal Investigator, MFM Consultant, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IND012018
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pre-Eclampsia
Keywords: Preeclampsia; Pravastatin; Maternal morbidity; Neonatal mortality; Neonatal morbidity
MeSH Terms: conditions — Pre-Eclampsia | interventions — Pravastatin

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Non Blinded Trial comparing low dose aspirin versus low dose aspirin and pravastatin in patients with high risk developing preeclampsia
Who Masked: Outcomes Assessor
Masking Description: The diagnosis is made by resident unaware of the medication patients received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pravastatin Treatment Group (Experimental): In this arm, the participant will be given aspirin 80 mg daily per oral and the study drugs, Pravastatin 2 x 20 mg per oral daily.
  Interventions: Drug: Pravastatin
- Control Group (No Intervention): In this arm, the participant will be given aspirin 80 mg daily per oral and the study drugs, Pravastatin 2 x 20 mg per oral daily.
  In this arm, the participant will be given aspirin 80 mg daily per oral, as it already a standard protocol for the high risk preeclampsia group

INTERVENTIONS:
Drug: Pravastatin — The participant will be given pravastatin 2 x 20 mg per oral daily
  Other Names: Pravastatin Sodium
  Arms: Pravastatin Treatment Group

SUMMARY:
BACKGROUND Preeclampsia is a major cause of maternal and neonatal morbidity worldwide. There is currently no cure for preeclampsia, the only definitive treatment is termination of pregnancy by induction of labour or caesarean section. Statin has been proposed to represent a new approach to improve disease outcome/prevent preeclampsia based on its multilayered activity toward pregnancy protection, including: protection of vascular endothelial cells survival, induce expression of heme oxygenase 1 (HO-1), inhibiting the release of soluble FMS-like tirosine kinase-1 (sFlt-1) and soluble endoglin (sEng), two main culprits in the pathophysiology of preeclampsia.

OBJECTIVE The aim of this study is to observe the effect of pravastatin administration in patients with high risk of preeclampsia in order to reduce maternal and neonatal mortality and morbidity.

METHODS This is a prospective randomized controlled clinical trial. The research will be held in 5 maternal fetal medicine centers in Indonesia (multicenter study). The recruitment will be done by permuted block random sampling methods, with sample size around 280 patients divides into two group. Patients with high risk of preeclampsia will be randomized either to get pravastatin 2 x 20 mg per oral and aspirin 1 x 80 mg (treatment group) or low dose aspirin only (control group). The patient will be followed regularly until delivery to obtain detailed maternal and neonatal outcome.

OUTCOME Primary Outcomes: Maternal preeclampsia, severe preeclampsia, gestational hypertension, indicated preterm delivery less than 37 weeks, indicated preterm delivery less than 34 weeks, maternal complications, length of hospital stay, and any serious adverse event.

Secondary Outcomes: Composite fetal/neonatal mortality and morbidity (stillbirth, neonatal death, respiratory distress syndrome, intracerebral hemorrhage, neonatal sepsis, intra uterine growth restriction [Small for Gestational Age (SGA) < 5th centile], and necrotizing enterocolitis), birthweight, birthweight percentile, level of care (well baby, intermediate, NICU), NICU length of stay, ventilator usage, and length of perinatal hospital stay.

KEYWORDS: pravastatin, preeclampsia, neonatal mortality, neonatal morbidity

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age 10 wk - 19 wk 6 day
* History of previous preeclampsia requiring birth < 37 weeks (risk 30%), or
* Patients with a combination of at least 2 major risk factors plus an abnormal uterine artery Doppler at 11-20 weeks gestation (risk preeclampsia 30%):

  * Major clinical risk factors (Obesity, strong family history of preeclampsia [mother or sister], maternal age > 40 years old, chronic hypertension, Policystic Ovarian Syndrome (PCOS), Chronic kidney disease, diabetes mellitus, multiple pregnancies, first pregnancy, pregnancy interval more than 10 years, new partner/husband, Reproductive technologies (IVF pregnancy), heritable thrombophilias, Booking Blood pressure >130/80 mmHg, family history of early onset cardiovascular disease, lower socioeconomic status)
  * Abnormal uterine artery Doppler defined as (Second trimester screening:

average resistance index > 0.58 and/or or early-diastolic diastolic notch. First trimester screening: Pulsatility index > 95th centile or PI > 1.5) or:

* First trimester screening (11+0 to 14+1 weeks): Combination of maternal risk factors, elevated MAP, and increased Uterine artery pulsatility index (UTPI).
* Second trimester screening (19+0 to 24+6 weeks): Combination of maternal risk factors, elevated MAP, and increased Uterine artery pulsatility index (UTPI).
* Combination of elevated mean arterial pressure (MAP > 90 mmHg) in the second trimester with abnormal uterine artery Doppler
* Combination elevated booking blood pressure (> 130/85 mmHg) with abnormal uterine artery Doppler
* Live fetus, no detectable fetal anomaly

Exclusion Criteria:

* Condition where the pregnancies should be terminated within 48 hours, on the basis of any indication (patients consume pravastatin less than 2 days).
* Contraindication to the statin use:

  * Hypersensitivity to pravastatin
  * Active liver disease
  * Pre pregnant renal insufficiency/kidney failure (history of hemodialysis)
* Current use of statin
* Participation in any other controlled trial of investigational medical products in pregnancy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | From date of randomization until date of delivery
  Including preeclampsia, preeclampsia with severe features, and gestational hypertension.
Preterm delivery | 20 - 34 weeks, and 34 - 37 weeks
  Including indicated preterm delivery < 34 weeks and < 37 weeks
Maternal complication | From date of randomization until date of delivery
  Any maternal complication caused by preeclampsia: eclampsia, seizure, HELLP syndrome, acute pulmonary edema, acute kidney injury, Cardivascular accident, liver failure, sepsis, and pneumonia

SECONDARY OUTCOMES:
Perinatal outcome | At delivery
  Gestational age at birth (days), birthweight (gram), birthweight percentile (INTERGROWTH), Apgar Score
Composite neonatal morbidity and mortality | At delivery
  stillbirths, neonatal death, respiratory distress syndrome, intracerebral hemorrhage, neonatal sepsis, necrotizing enterocolitis, length NICU admission, and length of stay

OTHER OUTCOMES:
The side effect of Pravastatin | Up to 6 month after birth
  Including adverse reactions, Serious Adverse Event (SAE), and Suspected Unexpected Serious Adverse Reaction (SUSAR)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ilham Aldika Akbar, MD, OBGYN, Principal Investigator — Universitas Airlangga
Locations (7):
- Indonesia (7):
  - Sanglah General Hospital, Denpasar, Bali
  - Dr. Moewardi Hospital, Surakarta, Central Java
  - Ramelan Naval Hospital, Surabaya, East Java
  - Dr. Soetomo Hospital, Surabaya, East Java
  - Adam Malik General Hospital, Medan, North Sumatra
  - Dr. Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi
  - Hasan Sadikin General Hospital, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed A, Ramma W. Unravelling the theories of pre-eclampsia: are the protective pathways the new paradigm? Br J Pharmacol. 2015 Mar;172(6):1574-86. doi: 10.1111/bph.12977. PMID 25303561
- [Background] Brennan LJ, Morton JS, Davidge ST. Vascular dysfunction in preeclampsia. Microcirculation. 2014 Jan;21(1):4-14. doi: 10.1111/micc.12079. PMID 23890192
- [Background] Cudmore M, Ahmad S, Al-Ani B, Fujisawa T, Coxall H, Chudasama K, Devey LR, Wigmore SJ, Abbas A, Hewett PW, Ahmed A. Negative regulation of soluble Flt-1 and soluble endoglin release by heme oxygenase-1. Circulation. 2007 Apr 3;115(13):1789-97. doi: 10.1161/CIRCULATIONAHA.106.660134. Epub 2007 Mar 26. PMID 17389265
- [Background] Costantine MM, Cleary K, Hebert MF, Ahmed MS, Brown LM, Ren Z, Easterling TR, Haas DM, Haneline LS, Caritis SN, Venkataramanan R, West H, D'Alton M, Hankins G; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric-Fetal Pharmacology Research Units Network. Safety and pharmacokinetics of pravastatin used for the prevention of preeclampsia in high-risk pregnant women: a pilot randomized controlled trial. Am J Obstet Gynecol. 2016 Jun;214(6):720.e1-720.e17. doi: 10.1016/j.ajog.2015.12.038. Epub 2015 Dec 23. PMID 26723196
- [Background] Ramma W, Ahmed A. Therapeutic potential of statins and the induction of heme oxygenase-1 in preeclampsia. J Reprod Immunol. 2014 Mar;101-102(100):153-160. doi: 10.1016/j.jri.2013.12.120. Epub 2014 Jan 16. PMID 24503248
- [Background] Ahmed A, Cudmore MJ. Can the biology of VEGF and haem oxygenases help solve pre-eclampsia? Biochem Soc Trans. 2009 Dec;37(Pt 6):1237-42. doi: 10.1042/BST0371237. PMID 19909254
- [Background] Dulak J, Deshane J, Jozkowicz A, Agarwal A. Heme oxygenase-1 and carbon monoxide in vascular pathobiology: focus on angiogenesis. Circulation. 2008 Jan 15;117(2):231-41. doi: 10.1161/CIRCULATIONAHA.107.698316. PMID 18195184
- [Background] Dekker G, Sibai B. Primary, secondary, and tertiary prevention of pre-eclampsia. Lancet. 2001 Jan 20;357(9251):209-15. doi: 10.1016/S0140-6736(00)03599-6. PMID 11213110
- [Background] Granger JP, Alexander BT, Llinas MT, Bennett WA, Khalil RA. Pathophysiology of hypertension during preeclampsia linking placental ischemia with endothelial dysfunction. Hypertension. 2001 Sep;38(3 Pt 2):718-22. doi: 10.1161/01.hyp.38.3.718. PMID 11566964
- [Background] Seki H. Balance of antiangiogenic and angiogenic factors in the context of the etiology of preeclampsia. Acta Obstet Gynecol Scand. 2014 Oct;93(10):959-64. doi: 10.1111/aogs.12473. Epub 2014 Sep 17. PMID 25139038
- [Background] Huppertz B. Placental origins of preeclampsia: challenging the current hypothesis. Hypertension. 2008 Apr;51(4):970-5. doi: 10.1161/HYPERTENSIONAHA.107.107607. Epub 2008 Feb 7. No abstract available. PMID 18259009
- [Background] Ofori B, Rey E, Berard A. Risk of congenital anomalies in pregnant users of statin drugs. Br J Clin Pharmacol. 2007 Oct;64(4):496-509. doi: 10.1111/j.1365-2125.2007.02905.x. Epub 2007 May 15. PMID 17506782
- [Background] Tranquilli AL, Dekker G, Magee L, Roberts J, Sibai BM, Steyn W, Zeeman GG, Brown MA. The classification, diagnosis and management of the hypertensive disorders of pregnancy: A revised statement from the ISSHP. Pregnancy Hypertens. 2014 Apr;4(2):97-104. doi: 10.1016/j.preghy.2014.02.001. Epub 2014 Feb 15. No abstract available. PMID 26104417
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Zarek J, Koren G. The fetal safety of statins: a systematic review and meta-analysis. J Obstet Gynaecol Can. 2014 Jun;36(6):506-509. doi: 10.1016/S1701-2163(15)30565-X. PMID 24927189
- [Background] von Dadelszen P, Magee LA. Pre-eclampsia: an update. Curr Hypertens Rep. 2014 Aug;16(8):454. doi: 10.1007/s11906-014-0454-8. PMID 24915961
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Maynard SE, Karumanchi SA. Angiogenic factors and preeclampsia. Semin Nephrol. 2011 Jan;31(1):33-46. doi: 10.1016/j.semnephrol.2010.10.004. PMID 21266263
- [Background] Hod T, Cerdeira AS, Karumanchi SA. Molecular Mechanisms of Preeclampsia. Cold Spring Harb Perspect Med. 2015 Aug 20;5(10):a023473. doi: 10.1101/cshperspect.a023473. PMID 26292986
- [Background] Teelucksingh S, El-Youssef J, Sohan K, Ramsewak S. Prolonged inadvertent pravastatin use in pregnancy. Reprod Toxicol. 2004 Mar-Apr;18(2):299-300. doi: 10.1016/j.reprotox.2003.11.003. No abstract available. PMID 15019727
- [Background] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK140561/ PMID 23741776